CLINICAL TRIAL: NCT05524727
Title: PEMOCS: Effects of a Concept-guided, PErsonalized, MOtor-Cognitive Training in Chronic Stroke - a RCT
Brief Title: PEMOCS: Personalized Motor-cognitive Training in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0614
Record Dates: First submitted 2022-08-02; First posted 2022-09-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: cognition; gait; mobility; training; chronic stroke; rehabilitation; virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Usual care + concept-guided, personalized, motor-cognitive training by means of an exergame
  Interventions: Other: Concept-guided, personalized, motor-cognitive training by means of an exergame
- Control Group (No Intervention): Usual care only

INTERVENTIONS:
Other: Concept-guided, personalized, motor-cognitive training by means of an exergame — 12 weeks, two times per week for 30-40min
  Arms: Intervention Group

SUMMARY:
In Switzerland, approximately 20'000 persons suffer a stroke each year. Despite carefully considered rehabilitation programs, full recovery is achieved only in a small proportion of stroke survivors (www.swissheart.ch). Studies suggest that motor-cognitive trainings can improve gait, balance, and mobility in chronic stoke survivors. However, little is known about the effect of motor-cognitive trainings on cognitive functioning in chronic stroke.

The aim of this study is to evaluate the effects of a motor-cognitive training added to usual care compared to usual care alone on cognitive functions, single- and dual-task mobility, gait and health-related quality of life.

In this single-blind RCT, 38 participants will be allocated randomly to either the intervention group (usual care + motor-cognitive training by means of an exergame for 12 weeks, 2x/week for 30-40 minutes) or the control group (usual care only). Both groups will attend three assessments, at baseline, post-intervention (12 weeks after baseline), and at follow-up (24 weeks after baseline). Global cognitive functioning will be the primary endpoint and a linear mixed model will be used for analysis.

Motor-cognitive trainings, especially exergames, bear the potential for further development of innovative long-term rehabilitation solutions for chronic stroke survivors. Cognitive deficits are a common unmet need restricting daily activities mentioned by chronic stroke survivors. Exergame training following personally tailored progression to generate optimal training load may help addressing this unmet need. Therefore, this study will contribute to the on-going research objective on how to improve the long-term care of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years) with chronic stroke (≥ 6 months post-stroke)
* Stroke: ischemic or haemorrhagic
* Able to stand for 3 minutes and walk 10 meters, functional ambulation category ≥ 3
* Able to follow a two-stage command
* Able to give informed consent as documented by signature

Exclusion Criteria:

* Unable or not willing to give informed consent
* Other neurological diseases (e.g. Parkinson's Disease, multiple sclerosis), except cognitive deficits or dementia
* Clinical contra-indications for the study intervention
* Unable to follow the study intervention or the test for the primary endpoint (MoCA), e.g. due to a neglect, aphasia or other language problems
* Overlapping enrolment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change of Montreal Cognitive Assessment Score | week 0, week 12 and week 24
  Widely used screening tool and cognitive outcome in neurological patients including stroke

SECONDARY OUTCOMES:
Change of Stroke Impact Scale 3.0 Score | week 0, week 12 and week 24
  Stroke-specific measurement tool assessing patient-reported health-related quality of life
Change of Simple Reaction Test Parameters | week 0, week 12 and week 24
  Widely used reliable and valid neuropsychological test assessing alertness
Change of Trail Making Test A & B Parameters | week 0, week 12 and week 24
  Widely used reliable and valid neuropsychological test assessing processing speed and executive functions
Change of Stroop Interference Test Parameters | week 0, week 12 and week 24
  Widely used reliable and valid neuropsychological test assessing the ability to inhibit the reaction to a more dominant stimulus in favour of the inquired reaction to a less dominant stimulus
Change of N-back test Parameters | week 0, week 12 and week 24
  Widely used reliable and valid neuropsychological test assessing working memory and related cognitive functions
Change of Mental Rotation Test Parameters | week 0, week 12 and week 24
  Measures the ability to mentally rotate abstract objects
Change in Single- and cognitive Dual-Task Timed Up and Go Test Parameters and motor/cognitive dual task costs | week 0, week 12 and week 24
  Widely used, reliable and valid test of mobility and dual-task ability in various populations including stroke.
Change of 10 meter walk test Gait Parameters | week 0, week 12 and week 24
  Widely used test to assess gait speed and spatiotemporal gait parameters.
Change of Outdoor Gait Parameters | week 0, week 12 and week 24
  Assesses walking endurance and spatiotemporal gait parameters under daily-life conditions.

OTHER OUTCOMES:
Compliance Rate | week 12
  attended sessions / offered sessions
Adherence Rate | week 12
  attended training time / offered training time
Perceived Motor-Cognitive Task Difficulty | twice per week, week 0-12
  visual analogue scale after each training session, based on cognitive load theory, scale from 1-9, where 9 symbolizes most difficult
Perceived Performance | twice per week, week 0-12
  visual analogue scale after each training session, performance item of the National Aeronautics and Space Administration - Task Load Index, scale from 0 to 20, where 20 symbolizes highest performance
Dose and Content of Usual Care | once per week, week 0-24
  according to weekly questionnaire, based on TIDIeR checklist
Amount and Intensity of General Physical and Cognitive Activity | once per week, week 0-24
  according to weekly questionnaire, based on TIDIeR checklist

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Ambulante Reha Triemli Zürich, Zurich
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Huber SK, Knols RH, Held JPO, Betschart M, Gartmann S, Nauer N, de Bruin ED. PEMOCS: effects of a concept-guided, PErsonalized, MOtor-Cognitive exergame training on cognitive functions and gait in chronic Stroke-a randomized, controlled trial. Front Aging Neurosci. 2025 Mar 13;17:1514594. doi: 10.3389/fnagi.2025.1514594. eCollection 2025. PMID 40182756
- [Derived] Huber SK, Knols RH, Held JPO, Betschart M, de Bruin ED. PEMOCS: Evaluating the effects of a concept-guided, PErsonalised, MOtor-Cognitive exergame training on cognitive functions and gait in chronic Stroke-study protocol for a randomised controlled trial. Trials. 2024 Jul 4;25(1):451. doi: 10.1186/s13063-024-08283-7. PMID 38965612